CLINICAL TRIAL: NCT01300507
Title: PREvention of Stent Thrombosis by an Interdisciplinary Global
Brief Title: PRESTIGE: PREvention of Stent Thrombosis by an Interdisciplinary Global European Effort
Acronym: PRESTIGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Deutsches Herzzentrum Muenchen (Other); European Union (Other)
Responsible Party: Principal Investigator, Prof Dr Walter Desmet, prof. dr. W. Desmet, KULeuven, Belgium and prof. T. Gerschlick, University Hospital Leicester, UK, University Hospitals Leuven, Belgium, University Hospital, Gasthuisberg
Other Study IDs: PRESTIGE 5.0 26.01.11
Record Dates: First submitted 2011-02-18; First posted 2011-02-21 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Coronary Artery Stent Thrombosis
Keywords: stent thrombosis; intra coronary imaging; blood platelet function testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimen: 1, thrombusaspiration from coronary arteries, storage and analysis at the German Heart Center Munich; 2, DNA-samples: storage at German Heart Center Munich, Antonius Hospital Nieuwegein, The Netherlands, University Hospitals Leuven Belgium and University Hospital Leicester, UK
Oversight: Data Monitoring Committee: No

SUMMARY:
The PRESTIGE-registry is a joint effort at 9 European heart centers to collect data regarding patients presenting with stent thrombosis in a dedicated database. There will be extensive clinical and procedural characterization, furthermore blood platelet function testing, intracoronary imaging, DNA-sampling and analysis of thrombus aspiration will be performed.

DETAILED DESCRIPTION:
Rationale: Stent Thrombosis (ST) is a serious complication of percutaneous coronary intervention (PCI) with stent implantation. Previous studies have been hampered by small sample size, in particular regarding the number of patients with late and very late ST and patients with DES thrombosis, and by incomplete patient characterisation, particularly concerning intracoronary imaging and blood platelet function data.

Objective: to identify novel predictors and to observe clinical outcome after an episode of ST, with the use of state-of-the-art new techniques such as OCT/IVUS, platelet function testing, genetic analysis.

Study design: multicenter matched case control study

Study population:

Cases: all patients presenting with definite ST. Expected number of patients to be included: 2000

Controls: patients undergoing PCI will be matched based on the following criteria:

Expected number of patients to be matched: 2000

1. who underwent a PCI for the same indication
2. who underwent a PCI on the same date (±5 days)
3. who underwent a PCI in the same interventional centre Main study parameters/endpoints: clinical, ECG, biochemical, angiographic, procedural, haematological, histopathological, genetic, OCT/IVUS-imaging, and follow-up characteristics Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Prior to PCI, 50 ml of whole blood will be drawn from all patients. Primary PCI for ST will be performed according to institutional best practise. During PCI, performance of Optical Coherence Tomography and/or Intravascular Ultrasound is encouraged. Thrombus aspiration is performed when indicated. During hospitalisation, all patients will be asked to fulfil a questionnaire regarding possible triggering mechanisms that might have provoked the ST. Patients will be asked to visit the patient clinic for platelet function 30 days after the acute phase of the ST. Finally, patients will be contacted for follow-up details.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting with stent thrombosis

Exclusion Criteria:

* patients refusing informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases: all patients presenting with definite ST. Expected number of patients to be included: 2000
  Controls: patients undergoing PCI will be matched based on the following criteria:
  Expected number of patients to be matched: 2000
  1. who underwent a PCI for the same indication
  2. who underwent a PCI on the same date (±5 days)
  3. who underwent a PCI in the same interventional centre
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2011-06; Primary Completion 2015-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
to identify novel factors responsible for the occurence of stent thrombosis | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Walter Desmet, MD, PhD, Principal Investigator — Dept. of Cardiology, University Hospitals Leuven, Belgium; Tony Gershlick, MD, PhD, Principal Investigator — Div. of Cardiology, Glenfield Hospital, Leicester, United Kingdom; Adnan Kastrati, MD, PhD, Study Chair — German Heart Institute, Munich, Germany; Steffen Massberg, MD, PhD, Study Chair — German Heart Institute, Munich, Germany; Tom Adriaenssens, MD, Study Director — Dept. of Cardiology, University Hospitals Leuven, Belgium; Wouter van Werkum, MD, PhD, Study Director — Dept. of Cardiology, St Antonius Hospital Nieuwegein, the Netherlands
Locations (1):
- UGasthuisberg, Leuven, Flemish Brabant, Belgium